CLINICAL TRIAL: NCT04332003
Title: A Randomized Controlled Double-Blind Multi-Center Clinical Trial Evaluating Remote Ischemic Conditioning (RIC) and Standard of Care vs. Sham Therapy and Standard Care in the Healing of Diabetic Foot Ulcers
Brief Title: Evaluating Remote Ischemic Conditioning (RIC) and Standard of Care vs. Sham Therapy and Standard Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: LifeCuff Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC-RIC
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: LifeCuff device includes a controller attached to a standard inflatable cuff used for blood pressure measurements.The controller includes a controller electronics board connected to a pneumatic assembly designed to automatically inflate and deflate the cuff to desired air pressures while monitoring and analyzing the oscillometric pulsations modulating the cuff pressure as captured by the system's pressure transducer. LifeCuff can be battery-powered or connected by an adaptor to a house electrical outlet.
Who Masked: Participant, Investigator
Masking Description: The subject and principle investigator will remain blinded throughout the trial. Every site will have a designated unblinded study coordinator. The unblinded coordinator will choose the appropriately labeled device for the subject during the weekly SOC visits. The patient will place the cuff and operate the device under the direction of the unblinded coordinator. The principle investigator is prohibited from entering the room during the treatment. The unblinded coordinator will place a sign on the outside of the study room door stating, "Do not enter. Study in Progress."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RIC Treatment (Active Comparator): Participants will receive active RIC treatment 3 times per week over the course of the study. Each session will last approximately 45 minutes
  Interventions: Device: Remote Ischemic Conditioning (RIC) Treatment
- SHAM Comparator (No Intervention): Participants will receive sham treatment 3 times per week over the course of the study. Each session will last approximately 45 minutes

INTERVENTIONS:
Device: Remote Ischemic Conditioning (RIC) Treatment — RIC treatment will be delivered by an automated device that delivers the RIC treatment (manufactured by LifeCuff Technologies).
  Arms: RIC Treatment

SUMMARY:
A double blind, randomized controlled clinical trial comparing wound closure rates of diabetic foot ulcers (DFUs) in subjects receiving active RIC treatment plus standard of care compared to those receiving sham treatment plus standard of care.

DETAILED DESCRIPTION:
The general objective of this double-blind study is to test the effectiveness of RIC in a population of patients with diabetic foot ulcers: Active treatment 3x per week (RIC) plus SOC compared to Sham Comparator 3x per week and SOC

Determine median time to initial wound closure in both active and sham group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of any gender between the ages of 18 and under 90 at the time of consent. The goal will be to enroll 50% of the subjects who are Medicare beneficiaries.
2. Target ulcer has a minimum area of 0.7 cm2 and a maximum area of 20.0 cm2, measured at randomization after sharp debridement, as assessed by photographic planimetry.
3. Target ulcer open for a minimum of 4 weeks and a maximum of 52 weeks duration prior to the screening visit.
4. Target ulcer is located on any aspect of the foot, including the toe, lateral dorsal, medial or plantar aspect of the foot. At least 50% of the ulcer must be below the malleolus.
5. Target ulcer is Wagner Grade I or Grade II without exposed bone.
6. Subjects' wound score on IDSA tool is Grade 1 or 2.
7. Adequate perfusion without critical limb ischemia, confirmed by vascular assessment of the affected foot through any of the following methods within 3 months of the first screening visit:

   Toe pressure ≥ 50 mm Hg; Ankle pressure ≥70 mm Hg; ABI between 0.7 and ≤ 1.3; TCOM ≥ 40 mmHg; Doppler ultrasound scan of peripheral blood flow with wave patterns that are triphasic or biphasic; Skin Perfusion Pressure (SPP) ≥30 mmHg.
8. Diagnosis of type 1 or 2 Diabetes mellitus,
9. Subject has a known glycated hemoglobin A1c (HbA1c) level of less than 12% within the last three months.
10. If subject has two or more ulcers, they must be separated by at least 2 cm and the largest one will be included as the study DFU though all will be similarly treated.
11. The target ulcer has been offloaded for at least 14 days prior to randomization.
12. Subject is willing to use prescribed off-loading method for the duration of the study.
13. Subject is available for the entire study period and all follow up visits. In addition, the subject is able and willing to adhere to the protocol requirements.
14. Subject able and willing to give written informed consent.

Exclusion Criteria:

1. Target ulcer is due to a non-diabetic etiology.
2. Presence in target ulcer of cellulitis, osteomyelitis or other clinical evidence of infection.
3. If the Target ulcer has reduced in area by 20% or more after 2 weeks of standard of care from the first screening visit (S1) to the TV-0/randomization visit.
4. An ulcer that has healed by more than 20% in the 2 weeks prior to screening: "historical" run-in period.
5. Presence of any foot ulcer (whether or not on the target foot) for which local or systemic antibiotic treatment is required.
6. A history of more than 8 weeks' treatment with immunosuppressants (including systemic corticosteroids at doses greater than 5mg of Prednisone or equivalent), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to initial screening, or treatments with such medications during the screening period, or anticipated requirement of such medications during the study.
7. Subjects with an amputation on the affected foot, only if it impedes proper offloading of the target DFU.
8. Subjects with active Charcot foot, or inactive Charcot foot, if it impedes proper offloading of the target DFU.
9. Women who are pregnant or considering becoming pregnant within the next 6 months.
10. Presence of subject having recent or current alcohol or drug abuse.
11. Subjects with severe kidney disease who are currently untreated or undergoing dialysis treatment.
12. Participation in another study involving treatment with an investigational product within the previous 30 days.
13. Any other medical or psychological conditions that, in the opinion of the Investigator, may make subject's participation unreliable or may interfere with study assessments.
14. There is a history of radiation to the target ulcer.
15. Subject has received HBO less than 30 days prior to screening.
16. Subject has received a cellular tissue product (CTP) less than 30 days prior to screening.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Time to complete wound closure. | 12-18 months
  Specifically, to determine the median time to initial wound closure in both the active treatment group and the sham treatment group

SECONDARY OUTCOMES:
Percentage of target wounds achieving closure | 12-week healing period
  The proportion of wounds that heal in a 12-week period
Percentage wound area reduction from TV-0 per week measured with digital planimetry and physical examination | 12- week
  The percentage of reduction in wound area from baseline
Change in DFU maximum depth in mm assessed by the Principal Investigator and documented by computer planimetry | 12 week
  The change in depth in mm over from baseline
Change in score of each domain on the CWIQ (Cardiff Wound Impact Questionnaire) | Day 0, 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Assess the change in daily quality of life
Change in pain regarding to the ulcer assessed using PEG (Pain, Enjoyment and General Activity) Scale | Day 0, 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Assess change in pain level
The percentage of time offloaded | Day 0, 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Offloading compliance with a prescribed offloading boot.
Change in skin sensitivity on the foot | Day 0, 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Assess change in skin sensitivity on the foot tested by performing standardized monofilament test over a standardized set of points on the foot
Percentage of time wearing the boot | Day 0, 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Compliance with a prescribed offloading boot
Change in Foot Infection | Day 0, 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Change in Foot Infection measured by the IDSA (Infectious Diseases Society of America) infection scale
Change in Wound Drainage | Day 0, 3 weeks, 6 weeks, 9 weeks, and 12 weeks
  Qualitatively assess the change in amount of drainage (low, moderate, heavy)
Change in oxygenation at the wound site | Day 0, 3 weeks, 6 weeks, 9 weeks and 12 weeks
  Assess change in oxygenation at the wound site using Near Infrared Reflectance Oximetry in a sub-group of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD,FACS, Principal Investigator — SerenaGroup, Inc.

IPD SHARING:
Plan to Share IPD: No